CLINICAL TRIAL: NCT04245995
Title: Quantification of Blood Loss Using a Novel Device in Comparison to Visually Estimated Blood Loss in a Simulated Blood Loss Scenario
Brief Title: Blood Loss Evaluation Using a Novel Device
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Florian Piekarski, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: KGU_FP_2020_CA1
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Blood Loss, Surgical; Transfusion; Patient Blood Management
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Feature Extraction Technology — The study´s aim was evaluation of the clinical applicability of the Feature Extraction Technology (FET) during a simulated blood loss scenario in comparison to visual estimation.

SUMMARY:
The study´s aim is to evaluate the clinical applicability of the Feature Extraction Technology (FET) during a simulated blood loss scenario.

DETAILED DESCRIPTION:
In an operating theatre blood loss will be simulated in different scenarios. Expired whole blood donations (provided by the German Red Cross, Institute of Transfusions Medicine, Goethe University Frankfurt) will be used. Blood will be diluted by full electrolyte solutions . Sponges and canisters will be prepared with a predetermined amount of blood.

Study participants will estimate total blood loss on sponges and canisters. Study members not knowing the correct amount of prepared blood will measure the blood loss in sponges and canisters by Feature Extraction Technology (FET) and by gravimetric method before and after estimation of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Health care professionals

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We include healthcare professionals.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | 02.05.2020 - 03.15.2020
  Visual versus novel device estimated blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Florian Piekarski, Dr. med., Principal Investigator — Goethe University, Frankfurt, Germany.
Locations (1):
- Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital Frankfurt, Goethe University, Frankfurt, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piekarski F, Gerdessen L, Schmitt E, Friedrichson B, Neef V, Meybohm P, Zacharowski K, Raimann FJ, Wunderer F. Quantification of Intraoperative Blood Loss in a Simulated Scenario Using a Novel Device. Shock. 2021 Jun 1;55(6):759-765. doi: 10.1097/SHK.0000000000001615. PMID 32694398